CLINICAL TRIAL: NCT03537807
Title: BHV-0223 Expanded Access Protocol in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Expanded Access Protocol of BHV-0223 for Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: No longer available | Type: Expanded Access
Sponsor: Biohaven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BHV0223-401
Record Dates: First submitted 2018-05-09; First posted 2018-05-25 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS; Lou Gehrig Disease; Lou Gehrig's Disease; Lou-Gehrigs Disease; Motor Neuron Disease, Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; ALS; Lou Gehrig Disease; Lou Gehrig's Disease; Lou-Gehrigs Disease; Motor Neuron Disease, Amyotrophic Lateral Sclerosis; Riluzole; Rilutek®; Sublingual; Oral formulation; Neuroprotective Agents; Administration, Sublingual; Administration, Oral; Biological Availability
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Riluzole

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Riluzole — For adult patients, one 40mg of BHV-0223, administered sublingually, on a twice daily basis (approximately every 12 hours).
  Other Names: Riluzole Zydis® sublingual

SUMMARY:
This is an open label expanded access protocol for the treatment of up to approximately 250 adult patients with amyotrophic lateral sclerosis (ALS) who have difficulty swallowing oral riluzole tablets and may be able to derive benefit from treatment with an alternative oral formulation of riluzole.

DETAILED DESCRIPTION:
Riluzole is indicated in the U.S. for the treatment of patients with amyotrophic lateral sclerosis (ALS). The commercially available dosage form is a 50mg oral tablet. This expanded access protocol (EAP) is designed to provide access to a dissolving tablet formulation of riluzole designed for sublingual (SL) administration, in patients with ALS who, in the opinion and clinical judgement of the treating physician, would benefit from treatment with BHV-0223.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed ALS of any type or duration
* Current or previous treatment with oral riluzole tablets, or patients who have never taken riluzole oral tablets, or patients who have successfully completed a clinical trial with BHV-0223 and were not withdrawn prematurely due to adverse events
* Swallowing difficulties, or patient or caregiver report choking one or more times per week, or investigator deems appropriate to treat with sublingual BHV-0223 because (s)he deems the patient cannot be satisfactorily treated with Rilutek®
* Adequate hepatic function

Exclusion Criteria:

* Patient with history of severe hypersensitivity reaction to riluzole oral tablets or BHV-0223
* Patient is known to have any other acute or chronic liver disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult